CLINICAL TRIAL: NCT06207981
Title: PRODIGE 85- KANALRAD : Prospective Randomized Phase III Study Evaluating Induction Chemotherapy (Modified DCF 4 Cycles) Followed by Chemoradiotherapy Compared to Standard Chemoradiotherapy for Locally Advanced Anal Squamous Cell Carcinoma (T3-4 or N1a, b or c)
Brief Title: Phase III Study Evaluating Induction Chemotherapy Followed by Chemoradiotherapy Compared to Standard Chemoradiotherapy for Locally Advanced SCCA
Acronym: KANALRAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Fondation ARCAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prodige 85 KANALRAD
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-02

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Induction Chemotherapy; Capecitabine; Mitomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): Pelvic chemoradiotherapy Radiotherapy consists of conformational intensity-modulated external irradiation with simultaneous integrated boost (IMRT-SIB) with 2 level of dose (30 sessions)
  * 49.5 Gy (5 x 1.65 Gy/week) to the pelvis
  * 60 Gy (5 x 2 Gy /week) to the primary tumor and initially involved nodes
  Concomitant Chemotherapy consists of Mitomycin-C (10 mg/m2 intravenous infusion at D1 and D29) and Capecitabine (1650 mg/m²/day divided in two oral intakes 825 mg/m² twice a day, five days a week). Patients should be counseled to only take capecitabine on the days when radiotherapy is being given
  Interventions: Drug: Concomitant chemotherapy (Capecitabin + Mitomycin-C); Radiation: radiotherapy
- Exeprimental arm (Experimental): Induction chemotherapy with mDCF (4 cycles) followed by pelvic chemoradiotherapy
  Induction chemotherapy consists of mDCF administered every 2 weeks:
  * Docetaxel (40 mg/m², day 1),
  * Cisplatin (40 mg/m², day 1)
  * 5-FU (1200 mg/m²/day IV for 2 days) Chemoradiotherapy is the same as described above in control arm
  Interventions: Drug: induction chemotherapy (mDCF); Drug: Concomitant chemotherapy (Capecitabin + Mitomycin-C); Radiation: radiotherapy

INTERVENTIONS:
Drug: induction chemotherapy (mDCF) — Induction chemotherapy consists of mDCF administered every 2 weeks:
  * Docetaxel (40 mg/m², day 1),
  * Cisplatin (40 mg/m², day 1)
  * 5-FU (1200 mg/m²/day IV for 2 days)
  Arms: Exeprimental arm
Drug: Concomitant chemotherapy (Capecitabin + Mitomycin-C) — Concomitant Chemotherapy consists of Mitomycin-C (10 mg/m2 intravenous infusion at D1 and D29) and Capecitabine (1650 mg/m²/day divided in two oral intakes 825 mg/m² twice a day, five days a week). Patients should be counseled to only take capecitabine on the days when radiotherapy is being given
Radiation: radiotherapy — Radiotherapy consists of conformational intensity-modulated external irradiation with simultaneous integrated boost (IMRT-SIB) with 2 level of dose (30 sessions)
  * 49.5 Gy (5 x 1.65 Gy/week) to the pelvis
  * 60 Gy (5 x 2 Gy /week) to the primary tumor and initially involved nodes

SUMMARY:
Squamous cell carcinoma of the anus is still a rare disease but its incidence increases mostly due to its association with human papillomavirus (HPV). When localized, the standard treatment combines radiotherapy and chemotherapy with 5FU and mitomycin-C. Chemoradiotherapy (CRT) achieves a good outcome for early stage tumors (T1-T2 tumors without nodal involvement), but more advanced tumors (T3-T4 or N1) are associated with a dismal prognosis. About 35 % of such patients relapse within two years after the end of treatment Recently, for metastatic or recurrent tumors after chemoradiotherapy, a chemotherapy combining docetaxel, cisplatin and 5FU (modified DCF protocol) has given very good results with a median overall survival of 39.2 months in 2 French trials (Epitopes HPV01 and 02). Our idea is to propose a new strategy , associating this chemotherapy (mDCF) followed by chemoradiotherapy to improve efficacy of the treatment for patients with locally advanced anal cancers. To this end, The principal investigator propose a national, multicenter, randomized phase 3 clinical trial to compare induction chemotherapy with mDCF followed by chemoradiotherapy versus standard chemoradiotherapy for locally advanced anal canal cancer.

the efficacy of the treatment will be evaluated by comparing disease-related event-free survival at 2 years according to the type of treatment. Other endpoints will also be evaluated such as overall survival and colostomy-free survival, treatment tolerability, response rate and quality of life.

This trial will be offered to patients over 18 years of age with locally advanced anal cancer without metastasis (T3-4 or N1). It is open to patients over 75 years of age subject to a favorable evaluation by an oncogeriatrician. It is also open to immunocompromised patients (HIV+) if their immunity is well controlled under antiretroviral treatment.The standard chemoradiotherapy treatment consists of 33 sessions of radiation, one session per day from Monday to Friday for 6.5 weeks. It is combined with chemotherapy that includes mitomycin during the first and fifth weeks of radiation therapy, as well as capecitabine that are taken on the days of radiation therapy.In the experimental arm, this chemoradiotherapy treatment is preceded by 4 sessions of mDCF chemotherapy performed every 2 weeks.After treatment, patients are followed up at 8 weeks, then every 4 months for 2 years, and every 6 months for the last year with clinical examination and imaging (CT and MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Anal Squamous cell carcinoma histologically proven
2. Locally advanced tumors without metastases

   * Stage T3 or T4
   * Stage N1 (a, b or c) - any T (T1 to T4)
3. Age ≥18 and ≤ 75 or > 75 in case of score G8 > 14 or favourable oncogeriatric assessment
4. Measurable tumor on MRI
5. Able to receive chemotherapy and radiotherapy
6. No major comorbidity that may preclude the delivery of treatment
7. Adequate hematologic function: absolute neutrophil count ≥ 1500/mm3, platelet count ≥ 100 000/mm3, Hb ≥ 9g/dl
8. Adequate renal function: creatinine clearance (according to MDRD formula) ≥ 60 ml/min
9. Adequate hepatic function: AST and ALT ≤ 2.5 × Upper Limit of Normal and total bilirubin ≤ 1.5 × ULN
10. WHO performance status < 2
11. Signature of informed consent
12. A negative pregnancy test for inclusion in the study for all female patients of child-bearing potential. In case of a "urine pregnancy test", it must be a highly sensitive urine pregnancy test, in accordance with the recommendations of the CTFG regarding pregnancy risk management (Recommendations related to contraception and pregnancy testing in clinical trials)
13. Female patients postmenopausal for at least one year or surgically infertile for at least 6 weeks, or effective contraception for male (until 6 months after the end of the investigational treatments) and female patients of childbearing potential (until 7.5 months after the end of treatment with cisplatine)
14. Patient to be covered by a regimen of French Social Security system.

Exclusion Criteria:

1. Presence of metastases
2. Stage T1N0 or T2N0
3. History of pelvic radiotherapy
4. Complete or partial Dihydropyrimidine dehydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL)
5. Positive HIV serology with CD4 < 400 / mm3
6. Presence of neuropathy > grade 2 according to NCIC-CTC 4.0
7. Contraindication for chemotherapy and/or radiotherapy
8. Concomitant treatment with CYP3A4 inhibitors or inducers
9. Symptomatic cardiac or coronary insufficiency
10. Progressive active infection or any unbalanced progressive severe condition in the last 6 months
11. No contraindication to MRI imaging
12. Other cancer treated within the last 3 years except in situ cervical carcinoma or basocellular/ spinocellular carcinoma or any other carcinoma in situ considered as cured
13. breastfeeding woman.
14. Persons deprived of liberty or under guardianship or incapable of giving consent
15. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.
16. Live attenuated vaccines within 4 weeks before randomization 17. In case of hearing problem 18. In case of combination with phenytoin with prophylactic aim 19. In case of recent or concomitant treatment brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-related event free survival (DREFS) at 2 years | 2 years after last patient completed treatment
  DREFS will be compared between the two arms . An event is defined as :progression, residual tumor at 6 months requiring APR, recurrence (local or metastatic) or death

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Vendrely, Md-pHD, Principal Investigator — University Hospital, Bordeaux
Locations (114):
- France (112):
  - AGEN-Cromg, Agen
  - Clinique Calabet, Agen
  - AIX EN PROVENCE CH Pays d'Aix, Aix-en-Provence
  - Amiens - Clinique de L'Europe, Amiens
  - ANTONY Hôpital Privé, Antony
  - Argenteuil - Ch, Argenteuil
  - ARRAS Les Bonnettes, Arras
  - ARRAS Marie Curie, Arras
  - AURILLAC-Henri Mondor, Aurillac
  - Centre Medico Chirurgical, Aurillac
  - AUXERRE CH GHT Unyon, Auxerre
  - Avignon Icap, Avignon
  - Avranches - Hopital Prive de La Baie, Avranches
  - Bayonne- Clinique Belharra, Bayonne
  - BEAUVAIS-Simone Veil, Beauvais
  - Besancon Chu, Besançon
  - Beuvry - Clinique Ambroise Pare, Beuvry
  - Beuvry Pierre Curie, Beuvry
  - Bordeaux - Privé - Tivoli, Bordeaux
  - BORDEAUX-Institut Bergonié, Bordeaux
  - Institut Bergonié, Bordeaux
  - Pessac - Chu -Haut Leveque, Bordeaux
  - Ch Duchenne, Boulogne-sur-Mer
  - BREST Pasteur Lanroze, Brest
  - CAEN Polyclinique du Parc, Caen
  - CAEN-François Baclesse, Caen
  - Cahors -Ch, Cahors
  - Caluire Et Cuire-Infirmerie Protestante, Caluire-et-Cuire
  - Chalon-Sur-Saone Hopital Sainte Marie, Chalon-sur-Saône
  - Chambery Ch, Chambéry
  - Chambray Les Tours-Roc37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Chu Estaing, Clermont-Ferrand
  - Centre de Radiothérapie Savoie Nord, Contamine-sur-Arve
  - Clinique de Flandre, Coudekerque-Branche
  - CRETEIL-Henri Mondor CHU, Créteil
  - DAX CH, Dax
  - DECHY-Léonard de Vinci, Dechy
  - Dijon - Chu François Mitterrand, Dijon
  - DIJON-GF Leclerc, Dijon
  - DIJON-Institut de Cancérologie de Bourgogne, Dijon
  - Ghm Grenoble - Institut Daniel Hollard, Grenoble
  - LA ROCHE-SUR-YON CHD Vendée, La Roche-sur-Yon
  - Guillaume Le Conquérant, Le Havre
  - LE HAVRE-l'Estuaire, Le Havre
  - LE MANS-CH Victor Hugo, Le Mans
  - Lille - Hopital Prive La Louviere, Lille
  - Limoges - Polyclinique Francois Chenieux, Limoges
  - Limoges-Chu Dupuytren, Limoges
  - LONGJUMEAU-GHNE Hôpital d'Antony, Longjumeau
  - Lorient - Groupe Hospitalier Bretagne Sud - Site Du Scorff, Lorient
  - LYON Jean Mermoz, Lyon
  - LYON- Léon Bérard, Lyon
  - LYON-Saint Joseph, Lyon
  - MARSEILLE Institut Paoli Calmettes, Marseille
  - MARSEILLE Saint-Joseph, Marseille
  - MARSEILLE-Hôpital la Timone, Marseille
  - Montbeliard Ch, Montbéliard
  - MONTPELLIER-ICM Val d'Aurelle, Montpellier
  - Mougins Cac, Mougins
  - MULHOUSE CH Emile Muller, Mulhouse
  - Nantes - Hopital Prive Du Confluent, Nantes
  - NEUILLY-SUR-SEINE GH Hartmann, Neuilly-sur-Seine
  - NICE-Antoine LACASSAGNE, Nice
  - Centre Hospitalier, Niort
  - Nimes Chu, Nîmes
  - ORLEANS Centre Hospitalier Régional, Orléans
  - OSNY-CHP Sainte-Marie, Osny
  - Paris - Ap-Hp - Hopital Tenon, Paris
  - Paris - Chu -Saint Louis Aphp, Paris
  - PARIS GHD Croix Saint-Simon, Paris
  - PARIS Hopital Europeen Georges-Pompidou, Paris
  - PARIS Institut Curie, Paris
  - PARIS-Saint Joseph, Paris
  - Pau Groupe de Radiotherapie Et D'Oncologie Des Pyrenees, Pau
  - PERIGUEUX-Hôpital Francheville, Périgueux
  - Plerin Hopital Prive Des Cotes D'Armor - Centre Cario, Plérin
  - POITIERS- CHU la Miletrie, Poitiers
  - PRINGY-Annecy Genevois CH, Pringy
  - REIMS-CHU Robert Debré, Reims
  - REIMS-Jean Godinot, Reims
  - Rennes - Centre Eugene Marquis, Rennes
  - Rennes Chu Pontchaillou, Rennes
  - RODEZ CH, Rodez
  - Hopitaux Prives Rouennais - Clinique Mathilde, Rouen
  - ROUEN-Frédéric Joliot, Rouen
  - Saint Denis Ch, Saint-Denis
  - CHU, Saint-Etienne
  - Saint Herblain Ico, Saint-Herblain
  - SAINT NAZAIRE CM l'Estuaire, Saint-Nazaire
  - Centre Hospitalier, Saint-Quentin
  - SARCELLES - Institut de Cancérologie Paris Nord, Sarcelles
  - Clinique Cote d'Emeraude, St-Malo
  - Saint Malo Ch, St-Malo
  - Strasbourg Icans, Strasbourg
  - STRASBOURG Sainte Anne, Strasbourg
  - Tarbes - Lourdes - Ch, Tarbes
  - Tarbes - Polyclinique de L'Ormeau, Tarbes
  - Thonon Les Bains - Hopitaux Du Leman, Thonon-les-Bains
  - Centre de Radiothérapie Saint-Louis, Toulon
  - TOULON-Sainte Anne, Toulon
  - Toulouse - Oncopole Institut Claudius Regaud, Toulouse
  - Toulouse Chu - Hopital Rangueil, Toulouse
  - TOULOUSE-Clinique Pasteur, Toulouse
  - TOURS CHU Trousseau, Tours
  - Valence - Centre Marie Curie, Valence
  - Valence Ch, Valence
  - VALENCE Drôme-Ardèche, Valence
  - Vandoeuvre Les Nancy-Ic Lorraine, Vandœuvre-lès-Nancy
  - VILLEJUIF Gustave Roussy, Villejuif
  - Centre de Radiothérapie Bayard, Villeurbanne
  - Villeurbanne Medipole Hopital Mutualiste Lyon, Villeurbanne
- Reunion (2):
  - Reunion - Chu Sud, Saint-Pierre
  - La Reunion - Clinique Prive Sainte Clotilde, Sainte-Clotilde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ffcd.fr/index.php?option=com_content&view=article&id=83&etude=00153&Itemid=144